CLINICAL TRIAL: NCT00223171
Title: Randomized, Multicentre, Phase III Study: Assessment of the Duration of Androgen Blockade Combined With Pelvic Irradiation in High-risk Prostate Cancers
Brief Title: Duration of Androgen Blockade Combined With Pelvic Irradiation in Prostate Cancers
Acronym: PCS IV
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Abdenour Nabid, Principal Investigator, Centre de recherche du Centre hospitalier universitaire de Sherbrooke
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DC-990-0056,1; DC-990-0056
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Prostate Cancer
Keywords: Stage T3 T4; PSA > 20; Gleason Score > 7
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 : 36 months AB + RT (Active Comparator): Androgen blockade : 36 months of androgen blockade : bicalutamide 50 mg die for one month, goserelin 10.8 mg x 12 Q 3 months + radiation therapy : pelvis 44 grays , prostate 70 grays (2 grays/fraction)
  Interventions: Drug: Androgen blockade + radiation therapy
- Arm 2 : 18 months AB + RT (Experimental): Androgen blockade 18 months : bicalutamide 50 mg die for one month, goserelin 10.8 mg x 6 Q 3 months + radiation therapy ( pelvis 44 grays , prostate 70 grays ,2 grays/fraction)
  Interventions: Drug: Androgen blockade + radiation therapy

INTERVENTIONS:
Drug: Androgen blockade + radiation therapy — Androgen blockade + radiation therapy

SUMMARY:
The objective of this study is to use as a reference the 36-month duration of hormonal therapy according to the European Organization for Research of the Treatment of Cancer (EORTC protocol 22863) : namely one-month of total androgen blockade followed by a luteinizing hormone releasing hormone (LHRH) agonist, all for three years, combined with pelvic and prostate irradiation; this arm is currently considered to be a standard for high-risk prostate cancers. The proposed study intends to challenge the duration of hormonal therapy and verify whether the five-year outcomes in favour of combined treatment in regard to survival (79% versus 62%) and local control (85% versus 48%) can be transposed for hormonal therapy that is half as long, namely 18 months, with the possibility of hormone salvage therapy in the event of biochemical and/or clinical failure (local, regional, or distant); this applies to both arms. The proposed study will compare survival in the two groups and evaluate in each one the total duration of initial hormonal therapy, followed by initial hormonal therapy combined with salvage hormonal therapy, the duration of salvage hormonal therapy until hormonal therapy resistance, and the side effects of this hormonal therapy, with everything being related to an assessment of the quality of life of these patients.

ELIGIBILITY:
Inclusion Criteria:

* To have at least one of the following three risk factors:

  * Tumour classified T3 or T4
  * Gleason score 8-10
  * Prostate-specific antigen (PSA) level > 20
* Performance status score of 0-1.
* Patients must sign a consent form before the start of the study.
* No evidence of regional disease: clinically negative regional adenopathies are revealed by imaging (computed axial tomography [CAT] scan, magnetic resonance imaging [MRI], lymphography) or surgical staging or negative pelvic node dissection.
* No distant metastasis. These patients must all have a negative bone scan 12 weeks prior to randomization.
* Hormonal therapy is allowed up to a maximum of two months before the consent form is signed, as long as the initial work-up was done, including having the requested deadlines respected.
* Patients with a previous history of cancer are eligible on the condition that they have not had any disease progression for more than five years.
* The patient must be available for treatments and follow-up visits.
* Treatments must start in the three weeks following randomization.

Exclusion Criteria:

* Severe medical or psychiatric problems that could compromise study compliance.
* Chronic hepatic disease, abnormal hepatic functions, i.e. aspartate aminotransferase, alanine aminotransferase > 1.5 times the upper normal limit.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 630 (Actual)
Dates: Start 2000-10; Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Specific survival | 10 years
Overall survival | 10 years
Treatment morbidity induced versus quality of life based on duration of hormonal therapy | 10 years

SECONDARY OUTCOMES:
Disease-free survival | 10 years
Site of tumour relapse | 10 years
Interval until first biochemical failure | 10 years
Interval until second biochemical failure during salvage androgen suppression (hormone-resistant tumour) | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Abdenour Nabid, MD, Principal Investigator — Centre de Recherche Clinique Étienne LeBel/CHUS Fleurimont
Locations (1):
- Centre de Recherche Clinique du CHUS, Sherbrooke, Quebec, Canada